CLINICAL TRIAL: NCT03633617
Title: A Phase 3, Randomized, 3-Part Study to Investigate the Efficacy and Safety of Dupilumab in Adult and Adolescent Patients With Eosinophilic Esophagitis (EoE)
Brief Title: Study to Determine the Efficacy and Safety of Dupilumab in Adult and Adolescent Patients With Eosinophilic Esophagitis (EoE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-EE-1774; 2018-000844-25 (EudraCT Number)
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Results first posted 2022-12-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Dupilumab or Placebo (Experimental): Part A consists of a 24-week double-blind treatment period. Participants will be randomized to receive dupilumab or placebo. At the end of the double-blind treatment visit (week 24), eligible participants may enter Part C. Participants who do not enter Part C will enter a 12-week follow-up period.
  Interventions: Drug: Dupilumab; Drug: Placebo
- Part B: Dupilumab or Placebo (Experimental): Part B consists of a 24-week double-blind treatment period. Participants will be randomized to receive dupilumab dosing regimen 1, dupilumab dosing regimen 2 or placebo. At the end of the double-blind treatment visit (week 24), eligible participants may enter Part C. Participants who do not enter Part C will enter a 12-week follow-up period.
  Interventions: Drug: Dupilumab; Drug: Placebo
- Part C: Dupilumab (Experimental): Part C is a 28-week extended active treatment period. Participants will receive dupilumab dosing regimen 1, dupilumab dosing regimen 2. At the end of the treatment period (week 52), participants will enter a 12-week follow-up period.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Solution for injection administered subcutaneously
  Other Names: DUPIXENT; REGN668; SAR231893
Drug: Placebo — Matching placebo
  Arms: Part A: Dupilumab or Placebo; Part B: Dupilumab or Placebo

SUMMARY:
The primary objectives of the study by study part are:

Part A:

To determine the treatment effect of dupilumab compared with placebo in adult and adolescent patients with EoE after 24 weeks of treatment as assessed by histological and clinical measures and to inform/confirm the final sample size determination for Part B.

Part B:

To demonstrate the efficacy of dupilumab treatment compared with placebo in adult and adolescent patients with EoE after 24 weeks of treatment as assessed by histological and clinical measures.

Part C:

To assess the safety and efficacy of dupilumab treatment in adult and adolescent patients with EoE after up to 52 weeks of treatment as assessed by histological and clinical measures.

The secondary objectives of the study are:

* To evaluate the safety, tolerability, and immunogenicity of dupilumab treatment for up to 52 weeks in adult and adolescent patients with EoE
* To explore the relationship between dupilumab concentration and responses in adult and adolescent patients with EoE, using descriptive analyses
* To evaluate the effects of dupilumab on transcriptomic signatures associated with EoE and type 2 inflammation
* To demonstrate the efficacy of dupilumab treatment compared to placebo after 24 weeks and 52 weeks of treatment in adult and adolescent patients with EoE who have previously received swallowed topical corticosteroids

ELIGIBILITY:
Key Inclusion Criteria (Parts A & B):

* A documented diagnosis of EoE by endoscopic biopsy
* Baseline endoscopic biopsies with a demonstration on central reading of intraepithelial eosinophilic infiltration
* History (by patient report) of an average of at least 2 episodes of dysphagia (with intake of solids) per week in the 4 weeks prior to screening

Key Exclusion Criteria (Parts A & B):

* Body weight ≤40 kg
* Prior participation in a dupilumab clinical trial, or past or current treatment with dupilumab
* Initiation or change of a food-elimination diet regimen or re-introduction of a previously eliminated food group in the 6 weeks prior to screening.
* Other causes of esophageal eosinophilia or the following conditions: hypereosinophilic syndrome and eosinophilic granulomatosis with polyangiitis (Churg-Strauss syndrome)
* Active Helicobacter pylori infection
* History of achalasia, Crohn's disease, ulcerative colitis, celiac disease, and prior esophageal surgery
* Any esophageal stricture unable to be passed with a standard, diagnostic, 9 to10 mm upper endoscope or any critical esophageal stricture that requires dilation at screening
* History of bleeding disorders or esophageal varices
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study

Key Exclusion Criteria (Part C):

* Participants who, during Part A or Part B, developed a serious adverse event (SAE) and/or adverse event (AE) deemed related to study drug, which in the opinion of the investigator could indicate that continued treatment with study drug may present an unreasonable risk for the participant
* Participants who became pregnant during Part A or Part B
* Participants who are prematurely discontinued from study drug due to an AE (patients who are prematurely discontinued from study drug due to lack of efficacy are eligible to enter Part C)
* Patients who did not undergo endoscopy with biopsies prior to receiving rescue treatment

Note: Other inclusion/ exclusion criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (90):
- United States (58):
  - Regeneron Study Site, Phoenix, Arizona
  - Regeneron Study Site, Scottsdale, Arizona
  - Regeneron Study Site, Little Rock, Arkansas
  - Regeneron Study Site, La Jolla, California
  - Regeneron Study Site, Los Angeles, California
  - Regeneron Study Site, Mountain View, California
  - Regeneron Study Site, Orange, California
  - Regeneron Study Site, Rolling Hills Estates, California
  - Regeneron Study Site, San Diego, California
  - Regeneron Study Site, Aurora, Colorado
  - Regeneron Study Site, Colorado Springs, Colorado
  - Regeneron Study Site, Lone Tree, Colorado
  - Regeneron Study Site, Bristol, Connecticut
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site, St. Petersburg, Florida
  - Regeneron Study Site, Boise, Idaho
  - Regeneron Study Site, Idaho Falls, Idaho
  - Regeneron Study Site #1, Chicago, Illinois
  - Regeneron Study Site #2, Chicago, Illinois
  - Regeneron Study Site, Park Ridge, Illinois
  - Regeneron Study Site, Urbana, Illinois
  - Regeneron Study Site, Indianapolis, Indiana
  - Regeneron Study Site, Clive, Iowa
  - Regeneron Study Site, Iowa City, Iowa
  - Regeneron Study Site, Topeka, Kansas
  - Regeneron Study Site, Hagerstown, Maryland
  - Regeneron Study Site, Boston, Massachusetts
  - Regeneron Study Site, Worcester, Massachusetts
  - Regeneron Study Site, Ann Arbor, Michigan
  - Regeneron Study Site, Chesterfield, Michigan
  - Regeneron Study Site, Plymouth, Minnesota
  - Regeneron Study Site, Rochester, Minnesota
  - Regeneron Study Site, Lincoln, Nebraska
  - Regeneron Study Site, Omaha, Nebraska
  - Regeneron Study Site, Great Neck, New York
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, The Bronx, New York
  - Regeneron Study Site, Chapel Hill, North Carolina
  - Regeneron Study Site, Cincinnati, Ohio
  - Regeneron Study Site, Dayton, Ohio
  - Regeneron Study Site, Dublin, Ohio
  - Regeneron Study Site, Mentor, Ohio
  - Regeneron Study Site, Hershey, Pennsylvania
  - Regeneron Study Site, Philadelphia, Pennsylvania
  - Regeneron Study Site, Charleston, South Carolina
  - Regeneron Study Site, Greenville, South Carolina
  - Regeneron Study Site, Johnson City, Tennessee
  - Regeneron Study Site, Memphis, Tennessee
  - Regeneron Study Site, Dallas, Texas
  - Regeneron Study Site, Fort Worth, Texas
  - Regeneron Study Site, Garland, Texas
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, San Antonio, Texas
  - Regeneron Study Site, Salt Lake City, Utah
  - Regeneron Study Site, Charlottesville, Virginia
  - Regeneron Study Site, Roanoke, Virginia
  - Regeneron Study Site, Seattle, Washington
  - Regeneron Study Site, Milwaukee, Wisconsin
- Australia (4):
  - Regeneron Study Site, Camperdown, New South Wales
  - Regeneron Study Site, Woolloongabba, Queensland
  - Regeneron Study Site, Elizabeth Vale, South Australia
  - Regeneron Study Site, Melbourne, Victoria
- Belgium (3):
  - Regeneron Study Site, Bruges
  - Regeneron Study Site, Edegem
  - Regeneron Study Site, Leuven
- Canada (4):
  - Regeneron Study Site, London, Ontario
  - Regeneron Study Site, Ottawa, Ontario
  - Regeneron Study Site, Montreal, Quebec
  - Regeneron Study Site, Hamilton
- France (2):
  - Regeneron Study Site, Pessac
  - Regeneron Study Site, Toulouse
- Germany (3):
  - Regeneron Study Site, Hanover
  - Regeneron Study Site, Magdeburg
  - Regeneron Study Site, Munich
- Italy (6):
  - Regeneron Study Site, Genoa
  - Regeneron Study Site, Milan
  - Regeneron Study Site, Naples
  - Regeneron Study Site, Pisa
  - Regeneron Study Site, Rome
  - Regeneron Study Site, Rozzano
- Netherlands (3):
  - Regeneron Study Site, Amsterdam
  - Regeneron Study Site, Maastricht
  - Regeneron Study Site, Nijmegen
- Spain (3):
  - Regeneron Study Site, Tomelloso, Ciudad Real
  - Regeneron Study Site, Barcelona
  - Regeneron Study Site, Madrid
- Regeneron Study Site, Stockholm, Sweden
- Regeneron Study Site, Zurich, Switzerland
- United Kingdom (2):
  - Regeneron Study Site, London, Whitechapel
  - Regeneron Study Site, Barnsley, Yorkshire

REFERENCES:
- [Derived] Bredenoord AJ, Dellon ES, Schlag C, Cianferoni A, Xia C, Pela T, Durrani S, Radwan A, Jacob-Nara JA. Dupilumab is efficacious for eosinophilic esophagitis irrespective of prior swallowed budesonide or fluticasone, or prior treatments used alongside swallowed topical corticosteroids: results from the phase 3, randomized, placebo-controlled, LIBERTY EoE TREET trial. Expert Rev Gastroenterol Hepatol. 2025 Jan-Feb;19(2):197-209. doi: 10.1080/17474124.2025.2461516. Epub 2025 Feb 5. PMID 39909733
- [Derived] Spergel JM, Chehade M, Dellon ES, Bredenoord AJ, Sun X, Glotfelty L, Shabbir A, Tilton ST, McCann E. Dupilumab Improves Health-Related Quality of Life and a Range of Symptoms in Patients With Eosinophilic Esophagitis. Am J Gastroenterol. 2024 Dec 1;119(12):2398-2407. doi: 10.14309/ajg.0000000000002924. Epub 2024 Jun 28. PMID 38940435
- [Derived] Bredenoord AJ, Dellon ES, Hirano I, Lucendo AJ, Schlag C, Sun X, Glotfelty L, Mannent L, Maloney J, Laws E, Mortensen E, Shabbir A. Dupilumab demonstrated efficacy and was well tolerated regardless of prior use of swallowed topical corticosteroids in adolescent and adult patients with eosinophilic oesophagitis: a subgroup analysis of the phase 3 LIBERTY EoE TREET study. Gut. 2024 Feb 23;73(3):398-406. doi: 10.1136/gutjnl-2023-330220. PMID 38050037
- [Derived] McCann E, Chehade M, Spergel JM, Yaworsky A, Symonds T, Stokes J, Tilton ST, Sun X, Kamat S. Validation of the novel Eosinophilic Esophagitis Impact Questionnaire. J Patient Rep Outcomes. 2023 Nov 27;7(1):120. doi: 10.1186/s41687-023-00654-z. PMID 38010430
- [Derived] Rothenberg ME, Dellon ES, Collins MH, Hirano I, Chehade M, Bredenoord AJ, Lucendo AJ, Spergel JM, Sun X, Hamilton JD, Mortensen E, Laws E, Maloney J, Mannent LP, McCann E, Liu X, Glotfelty L, Shabbir A. Efficacy and safety of dupilumab up to 52 weeks in adults and adolescents with eosinophilic oesophagitis (LIBERTY EoE TREET study): a multicentre, double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Gastroenterol Hepatol. 2023 Nov;8(11):990-1004. doi: 10.1016/S2468-1253(23)00204-2. Epub 2023 Aug 31. PMID 37660704
- [Derived] Dellon ES, Rothenberg ME, Collins MH, Hirano I, Chehade M, Bredenoord AJ, Lucendo AJ, Spergel JM, Aceves S, Sun X, Kosloski MP, Kamal MA, Hamilton JD, Beazley B, McCann E, Patel K, Mannent LP, Laws E, Akinlade B, Amin N, Lim WK, Wipperman MF, Ruddy M, Patel N, Weinreich DR, Yancopoulos GD, Shumel B, Maloney J, Giannelou A, Shabbir A. Dupilumab in Adults and Adolescents with Eosinophilic Esophagitis. N Engl J Med. 2022 Dec 22;387(25):2317-2330. doi: 10.1056/NEJMoa2205982. PMID 36546624

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A (24-week DBTP):157 participants screened, 81 randomized and received at least 1 dose of study drug; Part B (24-week DBTP): 462 participants screened, 240 randomized, 239 received treatment (1 participant randomized to placebo did not meet eligibility criteria and was discontinued prior to being treated).
Groups:
- Part A: Placebo: Participants received placebo matching dupilumab subcutaneously (SC) during Part A (a 24-week double-blind treatment period [DBTP]). At end of double-blind treatment visit, week 24 (one-week after last dose of study drug during the DBTP), eligible participants may enter into Part C. Participants who do not enter Part C will enter a 12-week follow-up period.
- Part A: Dupilumab 300 mg SC QW: Participants received dupilumab 300 milligrams (mg) SC once per week (QW) during Part A (a 24-week DBTP). At end of double-blind treatment visit, week 24 (one-week after last dose of study drug during the DBTP), eligible participants may enter into Part C. Participants who do not enter Part C will enter a 12-week follow-up period.
- Part B: Placebo: Participants received placebo matching dupilumab SC during Part B (a 24-week DBTP). At end of double-blind treatment visit, week 24 (one-week after last dose of study drug during the DBTP), eligible participants may enter into Part C. Participants who do not enter Part C will enter a 12-week follow-up period.
- Part B: Dupilumab 300 mg SC Q2W: Participants received dupilumab 300 mg once every 2 weeks (Q2W) SC during Part B (a 24-week DBTP). At end of double-blind treatment visit, week 24 (one-week after last dose of study drug during the DBTP), eligible participants may enter into Part C. Participants who do not enter Part C will enter a 12-week follow-up period.
- Part B: Dupilumab 300 mg SC QW: Participants received dupilumab 300 milligrams (mg) SC once per week (QW) during Part B (a 24-week DBTP). At end of double-blind treatment visit, week 24 (one-week after last dose of study drug during the DBTP), eligible participants may enter into Part C. Participants who do not enter Part C will enter a 12-week follow-up period.
- Part A/C: Placebo / Dupilumab 300 mg QW: Participants randomized to placebo in Part A, received dupilumab 300 mg QW for 28-week extended treatment (Part C) followed by 12-week follow-up. Participants who did not enter into Part C, entered follow-up.
- Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW: Participants randomized to dupilumab 300 mg QW in Part A continued to receive the same regimen for 28-week extended treatment (Part C) followed by 12-week follow-up. Participants who did not enter into Part C, entered follow-up.
- Part B/C: Placebo / Dupilumab 300 mg Q2W: Participants randomized to placebo in Part B were re-randomized in a 1:1 ratio to receive dupilumab 300 mg Q2W for 28-week extended treatment (Part C) followed by 12-week follow-up. Participants who did not enter into Part C, entered follow-up.
- Part B/C: Placebo / Dupilumab 300 mg QW: Participants randomized to placebo in Part B were re-randomized in a 1:1 ratio to receive dupilumab 300 mg QW for 28-week extended treatment (Part C) followed by 12-week follow-up. Participants who did not enter into Part C, entered follow-up.
- Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W: Participants randomized to dupilumab 300 mg Q2W in Part B continued to receive the same regimen for 28-week extended treatment (Part C) followed by 12-week follow-up. Participants who did not enter into Part C, entered follow-up.
- Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW: Participants randomized to dupilumab 300 mg QW during Part B, continued to receive the same regimen for 28-week extended treatment (Part C) followed by 12-week follow-up. Participants who did not enter into Part C, entered follow-up.
Period: Part A
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Started (Started Part A) | 39 | 42 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed week 24 visit for Part A) | 36 | 37 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Week 24 not performed due to Coronavirus Disease-2019 (COVID-19) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unconfirmed early termination visit | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Started (Started Part B (Participants from Part A were not eligible for Part B)) | 0 | 0 | 79 | 81 | 80 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed week 24 visit for Part B) | 0 | 0 | 74 | 79 | 75 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 5 | 2 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — COVID-19 Restrictions | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject randomized, but did not receive study drug; did not qualify for study | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C (& Follow-up)
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Started | 0 | 0 | 0 | 0 | 0 | 37 | 40 | 37 | 37 | 79 | 74
Completed Week 52 (End of Treatment) | 0 | 0 | 0 | 0 | 0 | 32 | 38 | 34 | 36 | 74 | 65
Completed (Completed follow-up (end of study)) | 0 | 0 | 0 | 0 | 0 | 30 | 35 | 33 | 36 | 67 | 64
Not Completed | 0 | 0 | 0 | 0 | 0 | 7 | 5 | 4 | 1 | 12 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 0 | 7 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — COVID-19 related | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Part A Full analysis set (FAS) includes all randomized participants in Part A; Part B FAS includes all randomized participants in Part B. Participants who participated in Part A were not eligible to participate in Part B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW | Total
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80 | 321
Age, Customized [Number; unit: Participants] — Part A: Age Population: Part A Full Analysis Set (FAS): All randomized participants in Part A
  Participants
    ≥ 12 to < 18 years old: number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    ≥ 12 to < 18 years old | 9 | 11 |  |  |  | 20
    ≥ 18 to < 40 years old: number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    ≥ 18 to < 40 years old | 22 | 13 |  |  |  | 35
    ≥ 40 to < 65 years old: number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    ≥ 40 to < 65 years old | 8 | 18 |  |  |  | 26
    ≥ 65 years old: number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    ≥ 65 years old | 0 | 0 |  |  |  | 0
Age, Customized [Number; unit: Participants] — Part B: Age Population: Part B FAS: All randomized participants in Part B
  Participants
    ≥ 12 to < 18 years old: number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    ≥ 12 to < 18 years old |  |  | 26 | 27 | 26 | 79
    ≥ 18 to < 40 years old: number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    ≥ 18 to < 40 years old |  |  | 38 | 35 | 38 | 111
    ≥ 40 to < 65 years old: number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    ≥ 40 to < 65 years old |  |  | 15 | 18 | 15 | 48
    ≥ 65 years old: number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    ≥ 65 years old |  |  | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Part A: Sex: Female, Male Population: Part A FAS: All randomized participants in Part A
  Participants
    number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    Female | 18 | 14 |  |  |  | 32
    Male | 21 | 28 |  |  |  | 49
Sex: Female, Male [Count of Participants; unit: Participants] — Part B: Sex: Female, Male Population: Part B FAS: All randomized participants in Part B
  Participants
    number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    Female |  |  | 21 | 36 | 30 | 87
    Male |  |  | 58 | 45 | 50 | 153
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Part A: Ethnicity (NIH/OMB) Population: Part A FAS: All randomized participants in Part A
  Participants
    number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    Hispanic or Latino | 1 | 4 |  |  |  | 5
    Not Hispanic or Latino | 38 | 38 |  |  |  | 76
    Unknown or Not Reported | 0 | 0 |  |  |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Part B: Ethnicity (NIH/OMB) Population: Part B FAS: All randomized participants in Part B
  Participants
    number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    Hispanic or Latino |  |  | 5 | 3 | 5 | 13
    Not Hispanic or Latino |  |  | 74 | 77 | 75 | 226
    Unknown or Not Reported |  |  | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants] — Part A: Race Population: Part A FAS: All randomized participants in Part A
  Participants
    White: number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    White | 37 | 41 |  |  |  | 78
    Black or African American: number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    Black or African American | 1 | 1 |  |  |  | 2
    Asian: number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    Asian | 0 | 0 |  |  |  | 0
    Other: number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    Other | 1 | 0 |  |  |  | 1
    Not reported: number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    Not reported | 0 | 0 |  |  |  | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Part B: Race Population: Part B FAS: All randomized participants in Part B
  Participants
    White: number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    White |  |  | 72 | 74 | 71 | 217
    Black or African American: number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    Black or African American |  |  | 3 | 3 | 2 | 8
    Asian: number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    Asian |  |  | 1 | 1 | 3 | 5
    Other: number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    Other |  |  | 2 | 2 | 3 | 7
    Not reported: number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    Not reported |  |  | 1 | 1 | 1 | 3
Part A: Dysphagia Symptom Questionnaire (DSQ) Total Score [Mean (Standard Deviation); unit: Score on a Scale] — The DSQ is used to measure the frequency and intensity of dysphagia. DSQ scores can range from 0 to 84, with a lower score indicating less-frequent or less-severe dysphagia. Population: Part A FAS: All randomized participants in Part A
  Score on a Scale
    number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    (all) | 35.1 (12.11) | 32.2 (12.66) |  |  |  | 33.6 (12.41)
Part B: Dysphagia Symptom Questionnaire (DSQ) Total Score [Mean (Standard Deviation); unit: Score on a Scale] — The DSQ is used to measure the frequency and intensity of dysphagia. DSQ scores can range from 0 to 84, with a lower score indicating less frequent or less severe dysphagia. Population: Part B FAS: All randomized participants in Part B
  Score on a Scale
    number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    (all) |  |  | 36.1 (10.55) | 35.6 (12.24) | 38.4 (10.70) | 36.7 (11.22)
Part A: Peak Eosinophils (eos) Count of Three Regions per High-power Field (/hpf) [Mean (Standard Deviation); unit: Eosinophils/high-power field (eos/hpf)] — Population: Part A FAS: All randomized participants in Part A
  Eosinophils/high-power field (eos/hpf)
    number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    (all) | 96.5 (54.69) | 82.6 (41.02) |  |  |  | 89.3 (48.29)
Part B: Peak Eosinophils (eos) Count of Three Regions per High-power Field (/hpf) [Mean (Standard Deviation); unit: Eosinophils/high-power field (eos/hpf)] — Population: Part B FAS: All randomized participants in Part B
  Eosinophils/high-power field (eos/hpf)
    number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    (all) |  |  | 84.3 (41.20) | 87.7 (49.37) | 89.2 (46.67) | 87.1 (45.76)
Part A: Eosinophilic Esophagitis (EoE) Histological Grade Calculated Mean Score (0 - 3) [Mean (Standard Deviation); unit: Score on a Scale] — Severity (grade) and extent (stage) of esophageal abnormalities were scored by blinded, central pathologists using a 4-point scale (0 normal; 3 maximum change) for eight features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells and lamina propria fibrosis (absent/present). Higher score indicates greater severity and extent of histological abnormalities. Population: Part A FAS: All randomized participants in Part A
  Score on a Scale
    number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    (all) | 1.324 (0.4676) | 1.260 (0.4088) |  |  |  | 1.291 (0.4365)
Part B: Eosinophilic Esophagitis (EoE) Histological Grade Calculated Mean Score (0 - 3) [Mean (Standard Deviation); unit: Score on a Scale] — Severity (grade) and extent (stage) of esophageal abnormalities were scored by blinded, central pathologists using a 4-point scale (0 normal; 3 maximum change) for eight features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells and lamina propria fibrosis (absent/present). Higher score indicates greater severity and extent of histological abnormalities. Population: Part B FAS: All randomized participants in Part B
  Score on a Scale
    number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    (all) |  |  | 1.226 (0.3996) | 1.245 (0.3721) | 1.305 (0.3882) | 1.259 (0.3865)
Part A: Eosinophilic Esophagitis (EoE) Histological Stage Calculated Mean Score (0 - 3) [Mean (Standard Deviation); unit: Score on a Scale] — Severity (grade) and extent (stage) of esophageal abnormalities were scored by blinded, central pathologists using a 4-point scale (0 normal; 3 maximum change) for eight features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells and lamina propria fibrosis (absent/present). Higher score indicates greater severity and extent of histological abnormalities. Population: Part A FAS: All randomized participants in Part A
  Score on a Scale
    number analyzed (Participants) | 39 | 42 | 0 | 0 | 0 | 81
    (all) | 1.376 (0.3972) | 1.299 (0.3334) |  |  |  | 1.336 (0.3653)
Part B: Eosinophilic Esophagitis (EoE) Histological Stage Calculated Mean Score (0 - 3) [Mean (Standard Deviation); unit: Score on a Scale] — Severity (grade) and extent (stage) of esophageal abnormalities were scored by blinded, central pathologists using a 4-point scale (0 normal; 3 maximum change) for eight features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells and lamina propria fibrosis (absent/present). Higher score indicates greater severity and extent of histological abnormalities. Population: Part B FAS: All randomized participants in Part B
  Score on a Scale
    number analyzed (Participants) | 0 | 0 | 79 | 81 | 80 | 240
    (all) |  |  | 1.216 (0.3608) | 1.248 (0.3182) | 1.294 (0.3256) | 1.253 (0.3353)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of ≤6 Eosinophils Per High-power Field (Eos/Hpf) in All Three Regions at Week 24
Description: Esophageal intraepithelial eosinophil count obtained by esophageal endoscopy with biopsies (all 3 esophageal regions: proximal, mid, and distal).
Time Frame: At week 24
Population: Part A Full Analysis Set (FAS): All participants randomized to Part A (Participants considered non-responder after rescue treatment use and multiple imputation (MI) method for missing due to COVID-19); Part B FAS: All participants randomized to Part B (Participants considered non-responder after rescue treatment use or missing not due to COVID-19 and MI method for missing or dosing interruption due to COVID-19)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Percentage of Participants | 5.1 [0.63 to 17.32] | 59.5 [43.28 to 74.37] | 6.3 [2.09 to 14.16] | 60.5 [49.01 to 71.19] | 58.8 [47.18 to 69.65]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in proportion = 55.3, 95% CI 2-sided [39.58 to 71.04] — Difference is dupilumab minus placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in proportion = 56.0, 95% CI 2-sided [43.44 to 68.54] — Difference is dupilumab minus placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in proportion = 53.5, 95% CI 2-sided [41.20 to 65.79] — Difference is dupilumab minus placebo

2. Primary Outcome: Absolute Change From Baseline in Dysphagia Symptom Questionnaire (DSQ) Total Score at Week 24
Description: The DSQ is used to measure the frequency and intensity of dysphagia. DSQ scores can range from 0 to 84, with a lower score indicating less-frequent or less-severe dysphagia.
Time Frame: Baseline and week 24
Population: Part A Full Analysis Set (FAS): All participant randomized to Part A (MI method with data set to missing after rescue treatment use); Part B FAS: All participants randomized to Part B (MI method with data set to missing after rescue treatment use)
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Score on a Scale | -9.60 [-15.056 to -4.136] | -21.92 [-26.870 to -16.967] | -13.86 [-17.605 to -10.120] | -14.37 [-18.018 to -10.723] | -23.78 [-27.427 to -20.131]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p = 0.0004, ANCOVA; LS Mean Difference = -12.32, 95% CI 2-sided [-19.107 to -5.537] — Dupilumab group vs. Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p = 0.8393, ANCOVA; LS Mean Difference = -0.51, 95% CI 2-sided [-5.423 to 4.406] — Dupilumab group vs. Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -9.92, 95% CI 2-sided [-14.811 to -5.022] — Dupilumab group vs. Placebo

3. Secondary Outcome: Percent Change From Baseline in Peak Esophageal Intraepithelial Eosinophil Count (Eos/Hpf) in All Three Regions at Week 24
Description: Esophageal intraepithelial eosinophil count obtained by esophageal endoscopy with biopsies (all 3 esophageal regions: proximal, mid, and distal). A greater esophageal intraepithelial eosinophil count from baseline indicates worsening disease.
Time Frame: Baseline and week 24
Population: Part A FAS (Worst-observation carried forward [WOCF]-MI method with data set to missing after rescue treatment use); Part B FAS (WOCF-MI method with WOCF for rescue treatment use and missing not due to COVID-19 and MI method for missing or dosing interruption due to COVID-19)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Change
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Percentage of Change | -2.98 [-17.886 to 11.921] | -71.24 [-84.863 to -57.613] | 8.38 [-11.677 to 28.433] | -70.84 [-87.095 to -54.585] | -80.24 [-96.589 to -63.895]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -68.26, 95% CI 2-sided [-86.896 to -49.615] — Dupilumab 300 mg QW vs Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -79.22, 95% CI 2-sided [-103.098 to -55.338] — Dupilumab 300 mg Q2W vs Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -88.62, 95% CI 2-sided [-112.194 to -65.046] — Dupilumab 300 mg QW vs Placebo

4. Secondary Outcome: Percent Change From Baseline in DSQ Total Score at Week 24
Description: as for outcome 2
Time Frame: Baseline and week 24
Population: Part A FAS (MI method with data set to missing after rescue treatment use); Part B FAS (MI method with data set to missing after rescue treatment use)
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Change
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Percentage of Change | -31.68 [-47.545 to -15.818] | -69.17 [-83.578 to -54.752] | -41.43 [-51.749 to -31.116] | -45.78 [-55.658 to -35.904] | -64.32 [-74.267 to 54.382]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -37.48, 95% CI 2-sided [-57.222 to -17.745] — Dupilumab 300 mg QW vs Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p = 0.5243, ANCOVA; LS Mean Difference = -4.35, 95% CI 2-sided [-17.734 to 9.038] — Dupilumab 300 mg Q2W vs Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p = 0.0008, ANCOVA; LS Mean Difference = -22.89, 95% CI 2-sided [-36.272 to -9.513] — Dupilumab 300 mg QW vs Placebo

5. Secondary Outcome: Absolute Change From Baseline in Eosinophilic Esophagitis Histology Scoring System (EoEHSS) Mean Grade Score at Week 24
Description: Severity (grade) and extent (stage) of esophageal abnormalities were scored by blinded, central pathologists using a 4-point scale (0 normal; 3 maximum change) for eight features: eosinophil density, basal zone hyperplasia, eosinophil abscesses, eosinophil surface layering, dilated intercellular spaces, surface epithelial alteration, dyskeratotic epithelial cells and lamina propria fibrosis (absent/present). Higher score indicates greater severity and extent of histological abnormalities.
Time Frame: Baseline and week 24
Population: Part A FAS (WOCF-MI method with data set to missing after rescue treatment use); Part B FAS (WOCF-MI method with WOCF for rescue treatment use and missing not due to COVID-19 and MI method for missing or dosing interruption due to COVID-19)
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Score on a Scale | -0.001 [-0.1166 to 0.1139] | -0.761 [-0.8732 to -0.6484] | -0.148 [-0.2379 to -0.0584] | -0.814 [-0.8958 to -0.7317] | -0.830 [-0.9136 to -0.7463]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.759, 95% CI 2-sided [-0.9061 to -0.6127] — Dupilumab 300 mg QW vs Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.666, 95% CI 2-sided [-0.7773 to -0.5538] — Dupilumab 300 mg Q2W vs Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.682, 95% CI 2-sided [-0.7929 to -0.5707] — Dupilumab 300 mg QW vs Placebo

6. Secondary Outcome: Absolute Change From Baseline in EoEHSS Mean Stage Score at Week 24
Description: as for outcome 5
Time Frame: Baseline and week 24
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Score on a Scale | -0.012 [-0.1243 to 0.0995] | -0.753 [-0.8627 to -0.6441] | -0.132 [-0.2179 to -0.0464] | -0.793 [-0.8713 to -0.7144] | -0.804 [-0.8839 to -0.7237]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.741, 95% CI 2-sided [-0.8842 to -0.5978] — Dupilumab 300 mg QW vs Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.661, 95% CI 2-sided [-0.7674 to -0.5540] — Dupilumab 300 mg Q2W vs Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.672, 95% CI 2-sided [-0.7778 to -0.5655] — Dupilumab 300 mg QW vs Placebo

7. Secondary Outcome: Absolute Change From Baseline in EoE Endoscopic Reference Total Score (EoE-EREFS) at Week 24
Description: EoE esophageal characteristics analyzed based on the EoE-EREFS, a scoring system for inflammatory and remodeling features of disease. The overall total score ranges from 0 to 18 with higher number indicating worse disease.
Time Frame: Baseline and week 24
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Score on a Scale | -0.3 [-1.11 to 0.50] | -3.2 [-3.98 to -2.38] | -0.6 [-1.37 to 0.12] | -4.6 [-5.24 to -3.89] | -4.5 [-5.17 to -3.77]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -2.9, 95% CI 2-sided [-3.91 to -1.84] — Dupilumab 300 mg QW vs Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -3.9, 95% CI 2-sided [-4.86 to -3.02] — Dupilumab 300 mg Q2W vs Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -3.8, 95% CI 2-sided [-4.77 to -2.93] — Dupilumab 300 mg QW vs Placebo

8. Secondary Outcome: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of <15 Eos/Hpf in All Three Regions at Week 24
Description: as for outcome 1
Time Frame: At week 24
Population: Part A FAS (Participants considered non-responder after rescue treatment use and MI method for missing due to COVID-19); Part B FAS (Participants considered non-responder after rescue treatment use or missing not due to COVID-19 and MI method for missing or dosing interruption due to COVID-19).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Percentage of Participants | 7.7 [1.62 to 20.87] | 64.3 [48.03 to 78.45] | 7.6 [2.84 to 15.80] | 79.0 [68.54 to 87.27] | 82.5 [72.38 to 90.09]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in proportion = 57.5, 95% CI 2-sided [41.69 to 73.33] — Difference is Dupilumab minus Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in proportion = 72.4, 95% CI 2-sided [61.05 to 83.70] — Difference is Dupilumab minus Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in proportion = 74.9, 95% CI 2-sided [64.25 to 85.50] — Difference is Dupilumab minus Placebo

9. Secondary Outcome: Normalized Enrichment Score (NES) for the Relative Change From Baseline in the EoE Diagnostic Panel (EDP) at Week 24
Description: NES reflects the degree to which the activity level of a set of disease transcripts is overrepresented at the extremes (top or bottom) of the entire ranked list of transcripts within a sample and is normalized by accounting for the number of transcripts in the set. An NES of 0 indicates no change from baseline, a negative score reflects a reduction in the disease score (more like normal) and a positive score reflects worsening (more active disease).
Time Frame: Baseline and week 24
Population: Part A FAS (Participants with NES Score in Part A; Last observation carried forward [LOCF] method with data set to missing after rescue treatment use); Part B FAS (Participants with NES Score in Part B; LOCF method with data set to missing after rescue treatment use)
Measure: Number; unit: Score on a Scale
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 29 | 31 | 41 | 44 | 40
Score on a Scale | -0.160 | -2.660 | -0.730 | -2.675 | -2.665
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Hodges-Lehmann estimator = -2.250, 95% CI 2-sided [-2.7200 to -1.7300] — Median Difference is Dupilumab minus Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Hodges-Lehmann estimator = -1.840, 95% CI 2-sided [-2.4200 to -1.1100] — Median Difference is Dupilumab minus Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Hodges-Lehmann estimator = -1.850, 95% CI 2-sided [-2.4400 to -1.1500] — Median Difference is Dupilumab minus Placebo

10. Secondary Outcome: NES for the Relative Change From Baseline in the Type 2 Inflammation Signature (T2INF) at Week 24
Description: as for outcome 9
Time Frame: Baseline and week 24
Population: Part A FAS (Participants with NES Score in Part A; LOCF Method with data set to missing after rescue treatment use); Part B FAS (Participants with NES Score in Part B; LOCF method with data set to missing after rescue treatment use)
Measure: Number; unit: Score on a Scale
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 29 | 31 | 41 | 44 | 40
Score on a Scale | -0.320 | -1.970 | -0.640 | -1.950 | -1.930
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Hodges-Lehmann estimator = -1.590, 95% CI 2-sided [-1.7400 to -1.2700] — Median Difference is Dupilumab minus Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Hodges-Lehmann estimator = -1.255, 95% CI 2-sided [-1.7300 to -1.0500] — Median Difference is Dupilumab minus Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test; Hodges-Lehmann estimator = -1.275, 95% CI 2-sided [-1.8200 to -1.0700] — Median Difference is Dupilumab minus Placebo

11. Secondary Outcome: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of ≤1 Eos/Hpf in All Three Regions at Week 24
Description: as for outcome 1
Time Frame: At week 24
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Percentage of Participants | 0.0 [0.00 to 9.03] | 21.4 [10.30 to 36.81] | 1.3 [0.03 to 6.85] | 27.2 [17.87 to 38.19] | 28.8 [19.18 to 39.95]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p = 0.0017, Cochran-Mantel-Haenszel; Difference in proportion = 21.9, 95% CI 2-sided [9.42 to 34.38] — Difference is Dupilumab minus Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in proportion = 27.6, 95% CI 2-sided [17.20 to 38.09] — Difference is Dupilumab minus Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in proportion = 28.9, 95% CI 2-sided [18.36 to 39.46] — Difference is Dupilumab minus Placebo

12. Secondary Outcome: Absolute Change From Baseline in Health-related Quality of Life (QoL) Average Score as Measured by EoE Impact Questionnaire (EoE-IQ) at Week 24
Description: The EoE-IQ measures impact of EoE on emotional, social, work & school, & sleep aspects. Participants were asked to respond to 11 questions based on experience living with EoE during past 7 days. Response to each item is on a 5-point scale (1=Not at all [impacted] 2=A little, 3=Somewhat, 4=Quite a bit, 5=Extremely [impacted]). The average score is the sum of non-missing responses divided by the number of items with non-missing responses. The average score can range from 1 to 5; a higher score is indicative of a more negative impact.
Time Frame: Baseline and week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Score on a Scale | -0.246 [-0.4659 to -0.0266] | -0.614 [-0.8140 to -0.4149] | -0.578 [-0.6977 to -0.4585] | -0.593 [-0.7152 to -0.4706] | -0.887 [-1.0050 to -0.7685]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p = 0.0077, ANCOVA; LS Mean Difference = -0.368, 95% CI 2-sided [-0.6388 to -0.0975] — Dupilumab group vs Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p = 0.8586, ANCOVA; LS Mean Difference = -0.015, 95% CI 2-sided [-0.1782 to 0.1485] — Dupilumab group vs. Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -0.309, 95% CI 2-sided [-0.4703 to -0.1471] — Dupilumab group vs. Placebo

13. Secondary Outcome: Absolute Change From Baseline in Severity of EoE Symptoms Other Than Dysphagia as Measured by EoE Symptom Questionnaire (EoE-SQ) at Week 24
Description: The EoE-SQ asks about symptoms that participants with EoE may have (chest pain, stomach pain, burning feeling in chest, food or liquid coming back up into throat, throwing up) during the past 7 days. Response to the severity of each symptom based on the worst experience in the past 7 days is on a scale of 0 to 10 (higher is worse). The EoE-SQ severity score is calculated as the sum of the severity scores from questions 1 to 3 (chest pain, stomach pain, burning feeling in chest), which could range from 0 to 30; a higher score is indicative of more severe symptoms.
Time Frame: Baseline and week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Score on a Scale | -3.9 [-5.46 to -2.31] | -5.8 [-7.24 to -4.44] | -4.0 [-5.16 to -2.80] | -4.5 [-5.59 to -3.32] | -5.4 [-6.60 to 4.27]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p = 0.0467, ANCOVA; LS Mean Difference = -2.0, 95% CI 2-sided [-3.87 to -0.03] — Dupilumab group vs. Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p = 0.5469, ANCOVA; LS Mean Difference = -0.5, 95% CI [-2.03 to 1.08] — Dupilumab group vs. Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p = 0.0718, ANCOVA; LS Mean Difference = -1.5, 95% CI 2-sided [-3.0 to 0.13] — Dupilumab group vs. Placebo

14. Secondary Outcome: Absolute Change From Baseline in Frequency of EoE Symptoms Other Than Dysphagia as Measured by EoE-SQ at Week 24
Description: The EoE-SQ asks about symptoms that participants with EoE may have (chest pain, stomach pain, burning feeling in chest, food or liquid coming back up into throat, throwing up) during the past 7 days. Response to the frequency of each symptom is on a 5-point scale (1 = 'Never', 2 = 'One day', 3 = ' 2-6 days', 4 = 'Once a day', 5 = 'More than once a day'). The EoE-SQ frequency score is calculated as the sum of the frequency scores from the 5 items which could range from 5 to 25; a higher score is indicative of higher frequency of symptoms.
Time Frame: Baseline and week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Score on a Scale | -1.7 [-2.67 to -0.71] | -3.4 [-4.29 to -2.53] | -2.6 [-3.25 to -1.87] | -3.0 [-3.69 to -2.36] | -3.9 [-4.61 to -3.25]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p = 0.0051, ANCOVA; LS Mean Difference = -1.7, 95% CI 2-sided [-2.93 to -0.52] — Dupilumab group vs. Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p = 0.3152, ANCOVA; LS Mean Difference = -0.5, 95% CI 2-sided [-1.38 to 0.44] — Dupilumab group vs. Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p = 0.0037, ANCOVA; LS Mean Difference = -1.4, 95% CI 2-sided [-2.30 to 0.45] — Dupilumab group vs. Placebo

15. Secondary Outcome: Percentage of Participants Who Received Rescue Treatment During the Placebo-controlled, Double-blind Treatment Period at Week 24
Time Frame: At week 24
Population: Part A FAS; Part B FAS
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 39 | 42 | 79 | 81 | 80
Percentage of Participants | 12.8 [4.30 to 27.43] | 0.0 [0.00 to 8.41] | 2.5 [0.31 to 8.85] | 1.2 [0.03 to 6.69] | 2.5 [0.30 to 8.74]
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Dupilumab 300 mg SC QW; Test type: Superiority; p = 0.0170, Cochran-Mantel-Haenszel; Difference in proportion = -12.7, 95% CI 2-sided [-23.21 to -2.26] — Difference is Dupilumab minus Placebo
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC Q2W; Test type: Superiority; p = 0.5493, Cochran-Mantel-Haenszel; Difference in proportion = -1.3, 95% CI 2-sided [-5.51 to 2.93] — Difference is Dupilumab minus Placebo
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: Dupilumab 300 mg SC QW; Test type: Superiority; p = 0.9887, Cochran-Mantel-Haenszel; Difference in proportion = 0.0, 95% CI 2-sided [-4.9 to 5.02] — Difference is Dupilumab minus Placebo

16. Secondary Outcome: Absolute Change From Baseline in Esophageal Distensibility Plateau Measured by Functional Lumen Imaging, if Collected, at Week 24
Time Frame: At week 24
Population: Due to only 7 participants in Part B with change from baseline at week 24 data available across 3 treatment groups, results are not reported to protect the confidentiality of the participants.
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of ≤6 Eosinophils Per High-power Field (Eos/Hpf) in All Three Regions at Week 52
Description: as for outcome 1
Time Frame: At week 52
Population: Part C safety analysis set (SAF): All participants who were randomized in Part A/B, entered Part C, and received any study drug in Part C.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 30 | 34 | 32 | 37 | 73 | 65
Percentage of Participants | 60.0 | 55.9 | 71.9 | 67.6 | 74.0 | 84.6

18. Secondary Outcome: Absolute Change in Dysphagia Symptom Questionnaire (DSQ) Total Score at Week 52
Description: as for outcome 2
Time Frame: Baseline (of previous study part) and week 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 23 | 29 | 27 | 24 | 52 | 54
Score on a Scale | -21.71 (17.143) | -23.44 (16.149) | -23.69 (13.737) | -27.25 (11.457) | -20.87 (16.387) | -30.26 (15.389)

19. Secondary Outcome: Percent Change in DSQ Total Score at Week 52
Description: as for outcome 2
Time Frame: Baseline (of previous study part) and week 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 23 | 29 | 27 | 24 | 52 | 54
Percentage of Change | -65.87 (49.705) | -75.93 (36.892) | -71.01 (37.256) | -78.13 (31.003) | -61.19 (44.447) | -80.74 (32.866)

20. Secondary Outcome: Absolute Change in EoE Endoscopic Reference Total Score (EoE-EREFS) at Week 52
Description: as for outcome 7
Time Frame: Baseline (of previous study part) and week 52
Population: as for outcome 17
Measure: Median (Standard Deviation); unit: Score on a Scale
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 30 | 35 | 31 | 37 | 73 | 63
Score on a Scale | -3.9 (2.74) | -4.1 (3.37) | -4.3 (3.21) | -6.1 (3.60) | -5.2 (3.40) | -5.3 (2.85)

21. Secondary Outcome: Percent Change in Peak Esophageal Intraepithelial Eosinophil Count (Eos/Hpf) in All Three Regions at Week 52
Description: as for outcome 3
Time Frame: Baseline (of previous study part) and week 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage of Change
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 30 | 34 | 32 | 37 | 73 | 65
Percentage of Change | -83.76 (24.996) | -88.59 (13.506) | -91.20 (13.037) | -84.21 (42.169) | -84.78 (40.973) | -95.85 (4.037)

22. Secondary Outcome: Absolute Change in EoE Histology Scoring System (EoEHSS) Mean Grade Score at Week 52
Description: as for outcome 5
Time Frame: Baseline (of previous study part) and week 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 30 | 34 | 32 | 37 | 73 | 65
Score on a Scale | -0.873 (0.5506) | -0.873 (0.3537) | -0.779 (0.4292) | -0.906 (0.3936) | -0.838 (0.4039) | -0.968 (0.4293)

23. Secondary Outcome: Absolute Change in EoEHSS Mean Stage Score at Week 52
Description: as for outcome 5
Time Frame: Baseline (of previous study part) and week 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 30 | 34 | 32 | 37 | 73 | 65
Score on a Scale | -0.874 (0.4630) | -0.891 (0.2770) | -0.710 (0.3783) | -0.871 (0.3510) | -0.809 (0.3434) | -0.932 (0.3730)

24. Secondary Outcome: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of <15 Eos/Hpf in All Three Regions at Week 52
Description: as for outcome 1
Time Frame: At week 52
Population: as for outcome 17
Measure: Number; unit: Percentage of Participants
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 30 | 34 | 32 | 37 | 73 | 65
Percentage of Participants | 70.0 | 82.4 | 87.5 | 78.4 | 83.6 | 100

25. Secondary Outcome: Percentage of Participants Achieving Peak Esophageal Intraepithelial Eosinophil Count of ≤1 Eos/Hpf in All Three Regions at Week 52
Description: as for outcome 1
Time Frame: At week 52
Population: as for outcome 17
Measure: Number; unit: Percentage of Participants
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 30 | 34 | 32 | 37 | 73 | 65
Percentage of Participants | 26.7 | 29.4 | 40.6 | 16.2 | 31.5 | 30.8

26. Secondary Outcome: Absolute Change in Health-related QOL as Measured by EoE-IQ at Week 52
Description: as for outcome 12
Time Frame: Baseline (of previous study part) and week 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 27 | 27 | 31 | 35 | 67 | 56
Score on a Scale | -0.954 (0.6690) | -0.911 (0.6344) | -1.021 (0.7169) | -0.858 (0.6360) | -0.773 (0.6217) | -0.935 (0.6883)

27. Secondary Outcome: Absolute Change From Baseline in Severity of EoE Symptoms Other Than Dysphagia as Measured by EoE-SQ at Week 52
Description: as for outcome 13
Time Frame: Baseline (of previous study part) and week 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 27 | 27 | 32 | 35 | 68 | 57
Score on a Scale | -7.2 (6.46) | -5.9 (6.80) | -6.2 (6.42) | -5.9 (6.47) | -4.7 (5.99) | -6.4 (6.86)

28. Secondary Outcome: Absolute Change From Baseline in Frequency of EoE Symptoms Other Than Dysphagia as Measured by EoE-SQ at Week 52
Description: as for outcome 14
Time Frame: Baseline (of previous study part) and week 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 27 | 27 | 32 | 35 | 68 | 57
Score on a Scale | -4.3 (3.78) | -3.2 (3.50) | -4.0 (3.54) | -3.8 (3.62) | -3.6 (3.45) | -4.7 (4.03)

29. Secondary Outcome: Percentage of Participants Who Received Rescue Medication During the 28-week Extended Active Treatment Period
Time Frame: Baseline (of Part C) to week 28
Measure: Number; unit: Percentage of Participants
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 37 | 40 | 37 | 37 | 79 | 74
Percentage of Participants | 8.1 | 0 | 2.7 | 2.7 | 0 | 1.4

30. Secondary Outcome: NES for the Relative Change From Baseline in EoE Diagnostic Panel (EDP) at Week 52
Description: as for outcome 9
Time Frame: Baseline (of previous study part) and week 52
Population: as for outcome 17
Measure: Median (Full Range); unit: Score on a Scale
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 27 | 30 | 17 | 24 | 60 | 49
Score on a Scale | -2.580 [-2.87 to -0.45] | -2.670 [-2.83 to -1.09] | -2.28 [-2.8 to -0.8] | -2.62 [-2.9 to -2.1] | -2.64 [-2.9 to 1.2] | -2.69 [-2.9 to -0.6]

31. Secondary Outcome: NES for the Relative Change in the Type 2 Inflammation Signature (T2INF) at Week 52
Description: as for outcome 9
Time Frame: Baseline (of previous study part) and week 52
Population: as for outcome 17
Measure: Median (Full Range); unit: Score on a Scale
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 27 | 30 | 17 | 24 | 60 | 49
Score on a Scale | -1.940 [-2.11 to -0.42] | -1.970 [-2.07 to -0.95] | -1.76 [-2.1 to -1.0] | -1.96 [-2.1 to -1.5] | -1.95 [-2.1 to 0.3] | -1.97 [-2.2 to -0.7]

32. Secondary Outcome: Concentration of Functional Dupilumab in Serum at Week 52
Time Frame: Baseline (of Part C) up to week 52
Population: The PK analysis set (PKAS) for Part A and Part C included all randomized participants who received any study drug and who had at least one non-missing drug concentration result following the first dose of study drug in the corresponding study part. The PKAS for Part B and Part C included all randomized participants who received any study drug and who had at least one non-missing drug concentration result following the first dose of study drug in the corresponding study part.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Arm/Group | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 34 | 38 | 36 | 37 | 77 | 69
milligrams per liter (mg/L)
  Week 32: number analyzed (Participants) | 28 | 24 | 31 | 35 | 71 | 58
  Week 32 | 101 (44.6) | 205 (76.8) | 46.0 (33.1) | 124 (56.7) | 74.0 (42.0) | 195 (94.6)
  Week 52: number analyzed (Participants) | 30 | 37 | 33 | 37 | 73 | 66
  Week 52 | 137 (81.6) | 152 (70.2) | 58.6 (36.5) | 151 (96.0) | 68.9 (45.7) | 176 (120)

33. Secondary Outcome: Incidence of Treatment-emergent Anti-drug Antibody (ADA) Response
Description: Number of treatment-emergent ADA responses to dupilumab reported.
Time Frame: Baseline (of previous study part) up to week 52
Population: ADA analysis set (AAS) Parts A & C: All participants who received any study drug & had at least 1 non-missing ADA result from dupilumab ADA assay after first dose of study drug in corresponding study part (according to treatment actually received); AAS Parts B & C: All participants who received any study drug & had at least 1 non-missing ADA result from dupilumab ADA assay after first dose of study drug in corresponding study part (according to treatment actually received).
Measure: Number; unit: Events
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg SC QW | Part B: Placebo | Part B: Dupilumab 300 mg SC Q2W | Part B: Dupilumab 300 mg SC QW | Part A/C: Placebo / Dupilumab 300 mg QW | Part A/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW | Part B/C: Placebo / Dupilumab 300 mg Q2W | Part B/C: Placebo / Dupilumab 300 mg QW | Part B/C: Dupilumab 300 mg Q2W / Dupilumab 300 mg Q2W | Part B/C: Dupilumab 300 mg QW / Dupilumab 300 mg QW
Number analyzed (Participants) | 39 | 42 | 77 | 77 | 76 | 35 | 39 | 36 | 37 | 77 | 69
Events | 0 | 0 | 0 | 2 | 1 | 4 | 1 | 1 | 0 | 5 | 0

ADVERSE EVENTS:
Time Frame: From day of first dose up to 12 weeks after end of treatment visit (week 52)
Groups:
- Part A: Placebo: Participants received placebo matching dupilumab SC during Part A (24-week DBTP). At end of week 24 visit (one-week after last dose of study drug during DBTP), eligible participants from Part A entered into 28-week extended treatment (Part C) and 12-week follow-up. Participants who did not enter into Part C, entered follow-up period.
- Part A: Dupilumab 300 mg QW: Participants received dupilumab 300 mg SC QW during Part A (24-week DBTP). At end of week 24 visit (one-week after last dose of study drug during DBTP), eligible participants from Part A entered into 28-week extended treatment (Part C) and 12-week follow-up. Participants who did not enter into Part C, entered follow-up period.
- Part B: Placebo: Participants received placebo matching dupilumab SC during Part B (24-week DBTP). At end of week 24 visit (one-week after last dose of study drug during DBTP), eligible participants from Part B entered into 28-week extended treatment (Part C) and 12-week follow-up. Participants who did not enter into Part C, entered follow-up period.
- Part B: Dupilumab 300 mg Q2W: Participants received dupilumab 300 mg Q2W SC during Part B (24-week DBTP). At end of week 24 visit (one-week after last dose of study drug during DBTP), eligible participants from Part B entered into 28-week extended treatment (Part C) and 12-week follow-up. Participants who did not enter into Part C, entered follow-up period.
- Part B: Dupilumab 300 mg QW: Participants received dupilumab 300 mg SC QW during Part B (24-week DBTP). At end of week 24 visit (one-week after last dose of study drug during DBTP), eligible participants from Part B entered into 28-week extended treatment (Part C) and 12-week follow-up. Participants who did not enter into Part C, entered follow-up period.
- Part C: Dupilumab 300 mg Q2W (Placebo in Part B): Participants randomized to placebo in Part B were re-randomized in a 1:1 ratio to receive dupilumab 300 mg Q2W for 28-week extended treatment (Part C) followed by 12-week follow-up. Participants who did not enter into Part C, entered follow-up.
- Part C: Dupilumab 300 mg QW (Placebo in Part A or B): Participants randomized to placebo in Part A, received dupilumab 300 mg QW for 28-week extended treatment (Part C) followed by 12-week follow-up. Participants who did not enter into Part C, entered follow-up. Participants randomized to placebo in Part B were re-randomized in a 1:1 ratio to receive dupilumab 300 mg Q2W for 28-week extended treatment (Part C) followed by 12-week follow-up. Participants who did not enter into Part C, entered follow-up.
- Part C: Dupilumab 300 mg Q2W (Part B Regimen Continued): Participants randomized to dupilumab 300 mg Q2W in Part B continued to receive the same regimen for 28-week extended treatment (Part C) followed by 12-week follow-up. Participants who did not enter into Part C, entered follow-up.
- Part C: Dupilumab 300 mg QW (Part A or B Regimen Continued): Participants randomized to dupilumab 300 mg QW in Part A continued to receive the same regimen for 28-week extended treatment (Part C) followed by 12-week follow-up. Participants who did not enter into Part C, entered follow-up. Participants randomized to dupilumab 300 mg QW during Part B, continued to receive the same regimen for 28-week extended treatment (Part C) followed by 12-week follow-up. Participants who did not enter into Part C, entered follow-up.
Arm/Group | Part A: Placebo | Part A: Dupilumab 300 mg QW | Part B: Placebo | Part B: Dupilumab 300 mg Q2W | Part B: Dupilumab 300 mg QW | Part C: Dupilumab 300 mg Q2W (Placebo in Part B) | Part C: Dupilumab 300 mg QW (Placebo in Part A or B) | Part C: Dupilumab 300 mg Q2W (Part B Regimen Continued) | Part C: Dupilumab 300 mg QW (Part A or B Regimen Continued)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/42 | 0/78 | 0/81 | 0/80 | 0/37 | 0/74 | 0/79 | 0/114
Serious Adverse Events (participants affected / at risk) | 2/39 | 2/42 | 1/78 | 2/81 | 5/80 | 1/37 | 3/74 | 1/79 | 4/114
Other Adverse Events (participants affected / at risk) | 28/39 | 26/42 | 41/78 | 57/81 | 50/80 | 19/37 | 44/74 | 47/79 | 62/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=39) | Part A: Dupilumab 300 mg QW (N=42) | Part B: Placebo (N=78) | Part B: Dupilumab 300 mg Q2W (N=81) | Part B: Dupilumab 300 mg QW (N=80) | Part C: Dupilumab 300 mg Q2W (Placebo in Part B) (N=37) | Part C: Dupilumab 300 mg QW (Placebo in Part A or B) (N=74) | Part C: Dupilumab 300 mg Q2W (Part B Regimen Continued) (N=79) | Part C: Dupilumab 300 mg QW (Part A or B Regimen Continued) (N=114)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Substance use disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Open globe injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Placebo (N=39) | Part A: Dupilumab 300 mg QW (N=42) | Part B: Placebo (N=78) | Part B: Dupilumab 300 mg Q2W (N=81) | Part B: Dupilumab 300 mg QW (N=80) | Part C: Dupilumab 300 mg Q2W (Placebo in Part B) (N=37) | Part C: Dupilumab 300 mg QW (Placebo in Part A or B) (N=74) | Part C: Dupilumab 300 mg Q2W (Part B Regimen Continued) (N=79) | Part C: Dupilumab 300 mg QW (Part A or B Regimen Continued) (N=114)
Injection site erythema (General disorders) | 6 (22) | 4 (12) | 9 (42) | 18 (93) | 8 (25) | 2 (32) | 6 (13) | 6 (36) | 10 (21)
Injection site reaction (General disorders) | 5 (19) | 9 (45) | 16 (69) | 18 (75) | 16 (84) | 3 (4) | 12 (40) | 14 (50) | 14 (101)
Injection site pain (General disorders) | 3 (6) | 5 (9) | 4 (21) | 10 (45) | 7 (39) | 4 (34) | 6 (7) | 6 (66) | 9 (45)
Injection site oedema (General disorders) | 2 (2) | 2 (7) | 3 (7) | 4 (4) | 0 (0) | 0 (0) | 3 (12) | 3 (12) | 3 (8)
Injection site pruritus (General disorders) | 2 (2) | 1 (1) | 3 (5) | 1 (6) | 4 (5) | 1 (6) | 1 (1) | 3 (8) | 0 (0)
Injection site bruising (General disorders) | 1 (2) | 1 (2) | 0 (0) | 6 (7) | 0 (0) | 1 (4) | 4 (4) | 1 (4) | 3 (3)
Injection site swelling (General disorders) | 1 (5) | 5 (7) | 2 (10) | 7 (12) | 10 (25) | 4 (4) | 0 (0) | 2 (4) | 4 (27)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 4 (20) | 2 (2) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 2 (4) | 6 (9) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 5 (6) | 3 (4) | 4 (5) | 2 (2) | 2 (2) | 7 (8) | 2 (3) | 5 (6)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 4 (4) | 1 (1) | 7 (7) | 8 (8) | 10 (10)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 6 (7)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 7 (9)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (2) | 7 (7) | 4 (4) | 5 (5) | 2 (3) | 1 (1) | 2 (2) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 4 (4) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 8 (12) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 4 (4) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (6) | 3 (5) | 3 (3) | 1 (1) | 3 (4) | 2 (2) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (9) | 2 (2) | 0 (0) | 0 (0) | 4 (6) | 2 (2) | 4 (6)
Headache (Nervous system disorders) | 4 (11) | 2 (7) | 9 (28) | 5 (10) | 7 (8) | 2 (6) | 4 (9) | 4 (6) | 5 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 6 (7) | 5 (6) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 4 (6) | 3 (3) | 2 (2) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 2 (2)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (3):
  • Study Protocol (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT03633617/Prot_000.pdf
  • Statistical Analysis Plan: Part A/Part C (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT03633617/SAP_001.pdf
  • Statistical Analysis Plan: Part B/Part C (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03633617/SAP_002.pdf